CLINICAL TRIAL: NCT04069715
Title: A Randomized, Placebo-controlled, Double-blind, Parallel Study to Determine the Effect of Farlong® NotoGinseng™ (Farlong® Ginseng Plus®) on Cholesterol and Blood Pressure
Brief Title: The Effect of Farlong® NotoGinseng™ (Ginseng Plus®) on Cholesterol and Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LongStar HealthPro, Inc. DBA Farlong Pharmaceutical (Industry)
Collaborators: Yunnan Panlong Yunhai Pharmaceutical Group Co., Ltd. (Industry); KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Farlong® NotoGinseng 16GCHY
Record Dates: First submitted 2017-08-30; First posted 2019-08-28 (Actual); Results first posted 2020-12-30 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Hyperlipidemias; Hypertension
Keywords: LDL-C; Blood pressure; triglycerides; HDL-C; total cholesterol; endothelial vasodilation; Hyperlipidemias; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension | interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: This was a randomized, placebo-controlled, double-blind, parallel study with a 4-week therapeutic lifestyle change diet (TLC) run-in period and a 12-week supplementation period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng) (Experimental): Participants will be instructed to take two capsules once per day in the morning, thirty minutes before a meal. Clinic staff will instruct participants to save all unused and open packages and return them to clinic at each subsequent visit (visit 3, visit 4 and visit 5) for a determination of compliance. If a dose is missed, participants are instructed to take one as soon as they remember that day. Participants will be advised not to exceed two capsules daily.
  Interventions: Dietary Supplement: Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng extract)
- Placebo (Placebo Comparator): Participants will be instructed to take two capsules once per day in the morning, thirty minutes before a meal. Clinic staff will instruct participants to save all unused and open packages and return them to clinic at each subsequent visit (visit 3, visit 4 and visit 5) for a determination of compliance. If a dose is missed, participants are instructed to take one as soon as they remember that day. Participants will be advised not to exceed two capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng extract) — A product made of highly concentrated pharmaceutical grade notoginseng root extract, and containing high potency bioactive components, notoginsenoside, ginsenoside Rb1, Rg1, Rd, Re and Rb2.
  Other Names: Farlong Panax NotoGinseng™; Notoginseng total saponins; Panax notoginseng saponins; Ginseng Plus®; Farlong Ginseng Plus®
  Arms: Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng)
Other: Placebo — Turmeric 0.4%, Rice Flour 76.6%, Magnesium stearate 23%, capsule shell (gelatin) 61 mg
  Arms: Placebo

SUMMARY:
In this randomized, placebo-controlled, double-blind parallel study in human participants with elevated LDL-C and elevated BP described here, the clinical benefits of Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng extract), a product made of highly concentrated pharmaceutical grade notoginseng root extract, and containing high potency bioactive components, notoginsenoside, ginsenoside Rb1 and ginsenoside Rg1, will be investigated for its efficacy on LDL-C and blood pressure.

DETAILED DESCRIPTION:
Health statistics include data on health disparities, global impact of cardiovascular diseases (CVDs) and risk factors including smoking, physical activity, body weight, cholesterol, blood sugar and blood pressure (BP) (1). Based on this, it is estimated that 33% of US adults had high blood pressure in 2009-2012 and during the same period, 43% of Americans had total cholesterol of 200 mg/dL or higher (2).

Chronic, elevated BP, defined as systolic BP (SBP) greater than 140 mmHg and diastolic BP (DBP) greater than 90 mmHg is clinically known as hypertension (3). Notably, hypertension is a strong, consistent, and independent risk factor for CVD and renal disease, including stroke, coronary heart disease, and kidney failure (4). Epidemiological evidence indicates that there is a log-linear relationship between elevated "bad" cholesterol, or low density lipoprotein-cholesterol (LDL-C) concentration, and relative risk of CVD (5). Lifestyle factors known to modify BP and cholesterol levels, including a balanced diet and exercise are not always met, highlighting the potential for nutritional supplementation.

The use of nutritional supplements, which might be effective in the reduction of high BP (hypertension) and hypercholesterolemia, is rapidly growing. However, most of the products available on the market have not been clinically evaluated for their effectiveness. Common ingredients found in cholesterol-lowering supplements include plant sterols. Plant sterols have been shown to reduce hypercholesterolemia in numerous experimental studies and in clinical trials, and are associated with lowering LDL-C by 10-15% (6;7). It has been estimated that consumption of at least 1.3 g of plant sterols/day may help to reduce the risk of heart disease by lowering blood cholesterol (8). Previous pre-clinical work reported that in addition to reduced cholesterol, supplementation with plant sterols can lower BP in hypertensive animals, although studies in humans are in early phases of development (9). Plant sterol supplementation may also improve vascular function, as one human trial found an association with sterol intake and lower levels of carotid wall thickness in older Amish participants (10).

Traditional Chinese Medicine has been used to treat cardiovascular diseases for thousands of years and species of the genus Panax plant are widely used in China and all over the world. Panax notoginseng (Burk.) F.H. Chen, is one of about 12 species in the Panax genus of the Araliaceae. Due to its sensitivity to light, P notoginseng is restricted to narrow geographic regions growing at an altitude of 1200-2000 m, primarily in the Wenshan mountains of Yunnan province in the People's Republic of China. The plant grows to a height of 30-60 cm and has dark green leaves branching from the stem where it typically bears a cluster of berries in the middle (11). The root of P notoginseng has a 400-year old history as a tonic and hemostatic drug; over 200 compounds have been isolated from this plant, exhibiting a variety of pharmacological effects, and appropriately enough the genus name "Panax" is derived from the Greek word (Pan = all + axos = medicine) meaning 'cure all' (12). Historically, Chinese medicine ascribes Panax ginseng C.A. Meyer to tonifying "qi", while P notoginseng nourishes the blood by dissipating blood stasis, inhibiting bleeding, enhancing circulation and alleviating pain. While the radix and rhizome of P notoginseng are used for bleeding disorders, the flower of this plant has been noted for several properties, including but not limited to, treating hypertension, and rejuvenating the liver (11). In the literature, extracts from P notoginseng have been referred to as Sanchitongshu, Xueshuantong, Sanqi or Tianqi and these ginsenosides from P notoginseng have collectively been referred to as Panax Notoginsenoside Saponins.

The primary bioactive ingredients in notoginseng plants are saponins, of which more than 60 have been identified (13). Saponins from notoginseng plant exert angiogenic effects by activating vascular endothelial growth factor and its receptor in downstream signaling pathways (14;15). Further, ginsenoside Rg5, a compound newly synthesized during the steaming process of notoginseng was found to promote angiogenesis and improve hypertension in animal models without adverse effects in the blood vasculature (16). Rg5 specifically increased phosphorylation of insulin-like growth factor-1 receptor (IGF-1R) resulting in stimulation of nitric oxide pathways to enhance angiogenesis (16). These studies suggest that notoginseng may have beneficial clinical applications in the management of CVD.

Currently, there is a lack of well-controlled trials evaluating the doses and effects of notoginseng (17). In this context, it is imperative to conduct well-controlled clinical trials that may unravel the mechanism (s) of action as well as evaluate the clinical potential of notoginseng as a natural health product and dietary supplement. In this randomized, placebo-controlled, double-blind parallel study in human participants with elevated LDL-C and elevated BP described here, the clinical benefits of Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng extract), a product made of highly concentrated pharmaceutical grade notoginseng root extract, and containing high potency bioactive components, notoginsenoside, ginsenoside Rb1 and ginsenoside Rg1, will be investigated for its efficacy on LDL-C and BP.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females age 18-75 years (inclusive)
2. BMI 23.0 to 32.5 kg/m2
3. Participants with LDL-C ≥2.6 mmol/L and <3.8 mmol/L (≥ 100 mg/dL and < 150 mg/dL)
4. Participants with pre-hypertension (systolic blood pressure of greater than or equal to 100 and less than 140 mmHg)
5. Participants agree to follow a therapeutic lifestyle changes (TLC) diet
6. If female, participant is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation)

   OR

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (DepoProvera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method (condoms with spermicide or diaphragm with spermicide)
   * Intrauterine devices
   * Vasectomy of partner (shown successful as per appropriate follow-up)
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
7. Willing to maintain current physical activity patterns throughout the study
8. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
9. Healthy as determined by laboratory results, medical history, and physical exam
10. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. History of allergic reaction or hypersensitivity to any of the study supplement components
2. Pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
3. Use of cholesterol-lowering or blood pressure lowering prescription drugs within the last 6 months prior to randomization
4. LDL-C ≥ 3.37 mmol/L (130 mg/dL), if the 10-year risk of cardiovascular event is ≥ 20% as estimated by the Framingham risk score
5. LDL-C > 3.5 mmol/L (135.34 mg/dL) OR if the total cholesterol vs. HDL-C ratio is > 5.0 OR hs-CRP > 2 mg/L in males > 50 years and females > 60 years, and if the 10-year Framingham risk score is 10-19%
6. Total cholesterol vs. HDL-C ratio > 6.0, if the 10-year Framingham risk score is < 10%
7. Use of ginseng-based drinks or products
8. Health supplements that affect blood pressure and cholesterol levels other than vitamins and minerals, such as plant sterols, omega-3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, licorice or other blood pressure and cholesterol lowering nonprescription supplements within 1 month of enrollment and during the study
9. Persons on medications listed in section 4.3
10. BMI > 32.5 kg/m2
11. Individuals with a history of coronary artery disease, previous myocardial infarction, peripheral vascular disease, atherosclerosis, diabetic men > 45 years old, and diabetic women > 50 years
12. Use of medicinal marijuana
13. History of chronic use of alcohol (> 2 drinks/day) over the past 6 months
14. Currently smoking ≥ 20 cigarettes/day
15. Use of systemic antibiotics, corticosteroids, androgens, or phenytoin, and HRT (HRTs are allowed if participant has been on a stable dose for at least 3 months and intends to maintain their dosage regimen).
16. Significant or untreated medical disorders including uncontrolled diabetes, recent myocardial ischemia or infarction, unstable angina, peripheral vascular diseases/bruits, uncontrolled thyroid dysfunction, renal failure and serious renal diseases, chronic active hepatitis, acute hepatitis, cirrhosis of liver, AIDS, malignancy, recent cerebrovascular disease and neurological disorders or significant psychiatric illness
17. Unstable medical conditions
18. History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, gastrointestinal, renal, pulmonary, hepatic or biliary disease, autoimmune disorders or cancer (evidence of active lesions, chemotherapy or surgery in the past year)
19. Anticoagulant/ antiplatelet medications; see section 4.3 for concomitant medications that are exclusionary
20. Immunocompromised individuals
21. History of hemoglobinopathies such as sickle cell anemia, thalassemia, or sideroblastic anemia
22. Individuals who have followed the Therapeutic Lifestyle Changes (TLC) diet within 12 weeks of screening
23. Recent surgery or will be undergoing surgery that may have an effect on the study in the opinion of the Qualified Investigator
24. Participation in a clinical research trial within 30 days prior to randomization.
25. History of eating disorders.
26. Clinically significant abnormal laboratory results at screening
27. Exercise greater than 24 km (15 miles)/week or 4,000 kcal/week
28. Cognitively impaired and/or who are unable to give informed consent
29. Plan to donate blood during the study or within 30 days of completing the study
30. Any additional underlying medical or psychiatric condition, clinical disorder or laboratory finding, which in the opinion of the Qualified Investigator may interfere with study objectives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Farlong NotoGinseng™: Farlong NotoGinseng™ (Treatment Group)
- Placebo: Placebo Group
Period: Overall Study
Arm/Group | Farlong NotoGinseng™ | Placebo
Started | 47 | 48
Completed | 42 | 43
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Farlong NotoGinseng™ | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.83 (12.65) | 49.96 (11.85) | 50.39 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 12 | 16 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Central American | 3 | 0 | 3
  Eastern European White | 4 | 2 | 6
  Middle Eastern | 2 | 1 | 3
  South American | 1 | 3 | 4
  South Asian | 1 | 0 | 1
  Western European White | 36 | 42 | 78
Region of Enrollment [Number; unit: participants]
  Canada | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Serum LDL-C From Baseline to Week 12 Between Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng Extract) and Placebo After 12 Weeks of Supplementation.
Description: The difference in serum LDL-C (mmol/L) from baseline to week 12 between Farlong NotoGinseng™ (Farlong Ginseng Plus® Panax Notoginseng extract) and placebo after 12 weeks of supplementation.
Time Frame: 12 weeks
Population: ITT Population. The analysis population takes into account participants that were withdrawn by the qualified investigator and those who were withdrawn at their own request.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 41 | 43
percentage of change | -0.07 (0.47) | -0.12 (0.54)

2. Secondary Outcome: 1. The Difference in Serum LDL-C From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 1. The difference in serum LDL-C (mmol/L) from baseline to week 8 between Farlong Notoginseng and placebo
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 42 | 44
percentage of change | -0.11 (0.55) | 0.01 (0.42)

3. Secondary Outcome: 2. The Difference in Blood Pressure From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 2. The difference in blood pressure (mmHg) from baseline to week 8 between Farlong Notoginseng and placebo
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 43 | 44
percentage of change
  Systolic Blood Pressure | -0.22 (7.95) | -0.46 (9.99)
  Diastolic Blood Pressure | -0.51 (5.95) | -0.39 (7.65)

4. Secondary Outcome: 3. The Difference in Blood Pressure From Baseline to Week 12 Between Farlong Notoginseng and Placebo
Description: 3. The difference in blood pressure (mmHg) from baseline to week 12 between Farlong Notoginseng and placebo
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 42 | 44
percentage of change
  Systolic Blood Pressure | -1.47 (8.10) | 1.23 (9.57)
  Diastolic Blood Pressure | -0.18 (5.17) | 1.08 (6.89)

5. Secondary Outcome: 4. The Difference in Triglycerides From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 4. The difference in triglycerides (mmol/L) from baseline to week 8 between Farlong Notoginseng and placebo
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 43 | 45
percentage of change | 0.05 (0.63) | -0.11 (0.53)

6. Secondary Outcome: 5. The Difference in Triglycerides From Baseline to Week 12 Between Farlong Notoginseng and Placebo
Description: 5. The difference in triglycerides (mmol/L) from baseline to week 12 between Farlong Notoginseng and placebo
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 42 | 44
percentage of change | -0.03 (0.58) | -0.05 (0.6)

7. Secondary Outcome: 6. The Difference in HDL-C From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 6. The difference in HDL-C (mmol/L) from baseline to week 8 between Farlong Notoginseng and placebo
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 43 | 45
percentage of change | 0.02 (0.24) | -0.02 (0.17)

8. Secondary Outcome: 7. The Difference in HDL-C From Baseline to Week 12 Between Farlong Notoginseng and Placebo
Description: 7. The difference in HDL-C (mmol/L) from baseline to week 12 between Farlong Notoginseng and placebo
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 42 | 44
percentage of change | 0.03 (0.19) | -0.02 (0.15)

9. Secondary Outcome: 8. The Difference in Total Cholesterol From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 8. The difference in total cholesterol from baseline to week 8 between Farlong Notoginseng and placebo
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 43 | 45
percentage of change | -0.06 (0.73) | -0.03 (0.57)

10. Secondary Outcome: 9. The Difference in Total Cholesterol From Baseline to Week 12 Between Farlong Notoginseng and Placebo
Description: 9. The difference in total cholesterol from baseline to week 12 between Farlong Notoginseng and placebo
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 42 | 44
percentage of change | -0.01 (0.64) | -0.13 (0.60)

11. Secondary Outcome: 10. The Difference in Endothelial Vasodilation, as Measured by the EndoPAT, From Baseline to Week 8 Between Farlong Notoginseng and Placebo
Description: 10. The difference in endothelial vasodilation (LnRHI), as measured by the EndoPAT, from baseline to week 8 between Farlong Notoginseng and placebo. The reactive hyperemia index (RHI) is a measure of endothelial function and LnRHI is a similar index after natural log transformation (Normal: LnRHI > 0.51 Abnormal: LnRHI ≤ 0.51). An increase in LnRHI is indicative of improvement in endothelial function.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 41 | 39
percentage of change | 0.00 (0.35) | 0.00 (0.28)

12. Secondary Outcome: 11. The Difference in Endothelial Vasodilation, as Measured by the EndoPAT, From Baseline to Week 12 Between Farlong Notoginseng and Placebo
Description: 11. The difference in endothelial vasodilation (LnRHI), as measured by the EndoPAT, from baseline to week 12 between Farlong Notoginseng and placebo. The reactive hyperemia index (RHI) is a measure of endothelial function and LnRHI is a similar index after natural log transformation (Normal: LnRHI > 0.51 Abnormal: LnRHI ≤ 0.51). An increase in LnRHI is indicative of improvement in endothelial function.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Farlong NotoGinseng™ | Placebo
Number analyzed (Participants) | 38 | 37
percentage of change | -0.04 (0.40) | -0.06 (0.30)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Farlong NotoGinseng™ | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 23/47 | 20/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Farlong NotoGinseng™ (N=47) | Placebo (N=48)
Dizziness (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Influenza like illness (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Psoriasis (Immune system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT04069715/Prot_SAP_000.pdf